CLINICAL TRIAL: NCT03224104
Title: Study of TG02 in Elderly Newly Diagnosed or Adult Relapsed Patients With Anaplastic Astrocytoma or Glioblastoma: A Phase Ib Study
Brief Title: Multi-kinase Inhibitor TG02 (TG02) in Elderly Newly Diagnosed or Adult Relapsed Patients With Anaplastic Astrocytoma or Glioblastoma.
Acronym: STEAM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1608-BTG; 2017-001029-42 (EudraCT Number); TG02-402 (Other: Tragara Pharmaceuticals, Inc.)
Record Dates: First submitted 2017-07-06; First posted 2017-07-21 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Astrocytoma, Grade III; Glioblastoma
Keywords: elderly; TG02; newly diagnosed; first relapse
MeSH Terms: conditions — Astrocytoma; Glioblastoma | interventions — 14-methyl-20-oxa-5,7,14,26-tetraazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8(27),9,11,16,21,23-decaene; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A - TG02 + RT (Experimental): Elderly patients with IDH1R132H-non mutant and MGMT promoter-unmethylated anaplastic astrocytoma or glioblastoma who will receive TG02 and radiation therapy.
  Interventions: Drug: TG02; Radiation: Radiation Therapy
- Group B - TG02 + TMZ (Experimental): Elderly patients with IDH1R132H-non mutant and MGMT promoter-methylated anaplastic astrocytoma or glioblastoma who will receive TG02 and temozolomide.
  Interventions: Drug: TG02; Drug: Temozolomide
- Group C - TG02 (Experimental): Patients initially diagnosed with anaplastic astrocytoma or glioblastoma at first relapse post TMZ/RT --> TMZ therapy who will receive TG02.
  Interventions: Drug: TG02

INTERVENTIONS:
Drug: TG02 — The initial cohorts of Groups A and B will receive TG02 at 200 mg on intermittent schedules in combination with either RT or TMZ. TG02 will be escalated to 250 mg if the dose decision criteria are met in the first cohort.
  The initial cohort in Group C will receive TG02 alone at 250 mg on intermittent schedules. It will be continued at this dose if feasible or decreased to 200 or 150 mg if not tolerated.
Radiation: Radiation Therapy — For group A standard involved-field hypofractionated RT will be administered at 39.9 Gy in 15 fractions of 2.66 Gy for 3 weeks
  Arms: Group A - TG02 + RT
Drug: Temozolomide — For group B TMZ will be given in the standard 28-day cycle regimen (150-200 mg/m2) for 5 days.
  Arms: Group B - TG02 + TMZ

SUMMARY:
This is a three parallel cohort, open-labeled, non-randomized, multicenter study. All three cohorts will enroll independently.

DETAILED DESCRIPTION:
Group A will be composed of newly-diagnosed, elderly patients with Isocitrate dehydrogenase 1 (IDH1) gene non mutant (IDH1R132H) and O-6-methylguanine-DNA methyltransferase (MGMT) promoter-unmethylated anaplastic astrocytoma or glioblastoma who will receive TG02 and radiotherapy (RT).

Group B will be composed of newly-diagnosed, elderly patients with IDH1R132H-non mutant and MGMT promoter-methylated anaplastic astrocytoma or glioblastoma who will receive TG02 and temozolomide.

For both Groups A and B, there will be a classical 3+3 dose escalation and an expansion phase in the study. Up to a total of 24 evaluable patients in Group A and up to a total of 12 evaluable patients in Group B (up to 36 evaluable patients for Groups A and B).

Group C patients will be composed of patients initially diagnosed with IDH1R132H-non-mutant anaplastic astrocytoma or glioblastoma at first relapse post TMZ/RT-->TMZ therapy who will receive TG02.

ELIGIBILITY:
Specifics for groups A and B

* Newly diagnosed glioblastoma or anaplastic astrocytoma, IDH1R132H-non-mutant by immunohistochemistry locally assessed, with formalin-fixed, paraffin-embedded (FFPE) tissue available for central MGMT testing and optional biomarker studies (treatment allocation will be performed based on centrally assessed MGMT result)
* Tumor debulking surgery, including partial resection
* Age > 65 and considered non-eligible for combination therapy (TMZ/RT→TMZ) in Investigator's opinion
* No prior RT with overlap of radiation fields with the planned RT in this study (Group A)
* No prior therapy for glioblastoma or anaplastic astrocytoma before surgery
* Brain MRI within 14 days before the first dose of TG02

Specifics for group C

* IDH1R132H-non-mutant glioblastoma or anaplastic astrocytoma at first relapse with tissue available from first surgery. [Per 2016 World Health Organization (WHO) classification, in patients older than 55 years of age at diagnosis with a histological diagnosis of glioblastoma, without a pre-existing lower grade glioma and with non-midline tumor location, immunohistochemical negativity for IDH1R132H suffices for classification as glioblastoma. In all other instances of diffuse gliomas, lack of IDH1R132H immunopositivity should be followed by IDH1 and isocitrate dehydrogenase 2 (IDH2) sequencing to detect or exclude other less common IDH mutations.]
* Brain MRI at the time of progression or 14 days before the first dose of TG02 and availability of last brain MRI before progression diagnosis for upload to the EORTC Imaging Platform for post-hoc central review of progression
* Diagnosis of recurrence more than 3 months after the end of RT for initial treatment
* Intention to be treated with standard TMZ/RT→TMZ for initial treatment (at least one dose of TMZ administered; RT alone or chemotherapy alone as initial treatment are not permitted)
* No discontinuation of TMZ for toxicity during first-line treatment
* No RT or stereotactic radiosurgery is allowed for the treatment of first recurrence prior to enrollment in this study
* Patient may have been operated for recurrence. If operated:
* surgery completed at least 2 weeks before initiation of TG02 and patients should have fully recovered as assessed by investigator. Criteria for full recovery include absence of active post-operative infection, recovery from medical complications (CTCAE grade 0 and 1 acceptable), and capacity for adequate fluid and food intake
* residual and measurable disease after surgery is not required but surgery must have confirmed the recurrence
* a post-surgery MRI should be available within 72 hours; the post-surgery MRI can be used as baseline if performed within 2 weeks prior to registration. If not, a baseline MRI has to be done within 2 weeks prior to registration
* For non-operated patients: recurrent disease must be at least one bi-dimensionally measurable contrast-enhancing lesion with clearly defined margins by MRI scan, with minimal diameters of 10 mm, visible on 2 or more axial slices 5 mm apart, based on a MRI scan done within 2 weeks prior to registration
* Age ≥ 18 years

All groups

* Karnofsky Performance Score (KPS) of 60-100
* Recovered from effects of debulking surgery, postoperative infection and other complications of surgery (if any) (CTCAE grade 0 and 1 acceptable)
* Adequate bone marrow, renal and hepatic function within the following ranges within 7 days before the first dose of TG02:
* white blood cell (WBC) ≥ 3 x109/L
* absolute neutrophil count (ANC) ≥ 1.5x109/L
* Platelet count of ≥ 100 x109/L independent of transfusion
* Hemoglobin ≥ 10 g/dl or ≥ 6.2 mmol/L
* Bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Cockcroft-Gault calculated or measured creatinine clearance of ≥ 30 mL/min
* No use of enzyme-inducing anti-epileptic drugs (EI-AED) within 7 days prior to the first dose of TG02
* Life expectancy > 8 weeks
* No history of ventricular arrhythmia or symptomatic conduction abnormality in past 12 months prior to registration
* No congestive heart failure (New York Heart Association Class III to IV, see Appendix C), symptomatic ischemia, uncontrolled by conventional intervention, or myocardial infarction within 6 months prior to enrollment
* No 12-lead ECG with a prolonged corrected QT interval (QTc) interval (males: > 450 ms; females: > 470 ms) as calculated by the Fridericia correction formula despite balancing of electrolytes at registration and/or discontinuing any drugs (for a time period corresponding to 5 half-lives) known to prolong QTc interval
* No known contraindication to imaging tracer or any product of contrast media
* No MRI contraindications
* No concurrent severe or uncontrolled medical disease (e.g., active systemic infection, diabetes, hypertension, coronary artery disease) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study
* No known human immunodeficiency virus infection or acquired immune deficiency syndrome
* No previous other malignancies, except for any previous malignancy which was treated with curative intent more than 3 years prior to enrollment, or adequately controlled limited basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix
* No pregnant women. Negative serum or urine pregnancy test within 72 hours prior to the first dose for women of childbearing potential (WOCBP). Nursing must be discontinued at least 1 hour before first dose.
* For men of reproductive potential and WOCBP, adequate contraception must be used throughout the study and for 6 months thereafter. For this study, acceptable methods of contraception include a reliable intrauterine device or a spermicide in combination with a barrier method. Hormonal forms of birth control (oral, implantable, or injectable) may only be used if combined with another highly effective form of birth control such as a spermicide combined with a barrier method
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments
* Ability to take oral medication
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration, written informed consent must be given according to International Conference on Harmonization ICH) / Good Clinical Practice (GCP), and national/local regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Le Rhun, Principal Investigator — CHRU de Lille
Locations (10):
- Universitaetskliniken der Uni Wien - Universitaetsklinikum Wien - AKH uniklinieken, Vienna, Austria
- France (3):
  - CHU de Lyon - CHU Lyon - Hopital neurologique Pierre Wertheimer, Bron
  - CHRU de Lille, Lille
  - Assistance Publique - Hopitaux de Marseille - Hôpital de La Timone, Marseille
- Germany (4):
  - Universitaetsklinikum Bonn, Bonn
  - Klinikum Der J.W. Goethe Universitaet-Klinik und Poliklinik fur Neurochirurgie, Frankfurt
  - Universitaetsklinikum Heidelberg - UniversitaetsKlinikum Heidelberg - Head Hospital, Heidelberg
  - Universitaetskliniken Regensburg - Universitaetsklinikum Regensburg, Regensburg
- Erasmus MC Cancer Institute - location Daniel den Hoed, Rotterdam, Netherlands
- UniversitaetsSpital Zurich, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient registration/enrollment was only accepted from authorized investigators. Patients were registered/enrolled on the EORTC online randomized trials access. After registration and shipment of sample has been done, the central laboratory assessed the o6-methylguanine-DNA-methyltransferase (MGMT) promoter methylation status. Based on the MGMT results, patients were allocated to group A or B. In group C, patients were directly enrolled.
Pre-assignment Details: In all 3 study groups, only eligible patients were enrolled.
Groups:
- Group A - TG02 + Radiotherapy (RT) Dose 1 100 mg; Group A - TG02 + Radiotherapy (RT) Dose 2 150 mg: Newly-diagnosed elderly patients (≥65 years) with IDH1R132H-non mutant and MGMT promoter-unmethylated brain tumors received TG02 orally twice weekly with radiation therapy (RT). TG02 was given on specific days of a 28-day cycle, and RT was administered at 40 Gy over 3 weeks. After combination therapy, patients received maintenance TG02 for up to 12 cycles or until disease progression. The dose of TG02 was escalated from 100 mg to 150 mg based on the occurrence of dose-limiting toxicities (DLTs) in cohorts of patients. If no or only one patient experienced a DLT at 150 mg, it was considered the maximum tolerated dose (MTD). If more than one patient experienced a DLT at either dose, the arm was closed. Patients without DLTs continued at the same dose unless severe side effects required adjustments.
- Group B - TG02 + Temozolomide (TMZ) Dose 1 100 mg; Group B - TG02 + Temozolomide (TMZ) Dose 2 150 mg: Elderly patients with IDH1R132H-non mutant and MGMT promoter-methylated tumors brain tumors received TG02 and temozolomide (TMZ). TG02 was taken on a schedule that varied in the first cycle but was consistent in subsequent cycles. TMZ was given in a standard 28-day cycle. Treatment continued until disease progression or for up to 12 cycles. After 12 cycles, patients could continue on the combination or single-agent TG02. The dose escalation for TG02 involved starting at 100 mg, with rules for escalating to 150 mg based on the occurrence of dose-limiting toxicities (DLTs). If certain numbers of patients experienced DLTs, the dose would not be escalated, or the arm might be closed. Patients without DLTs continued at the same dose unless a severe side effect required a dose adjustment.
- Group C - TG02: Anaplastic Astrocytoma (AA) and Glioblastoma (GBM) patients at first relapse after TMZ/RT followed by maintenance TMZ therapy will receive single agent TG02 at 150 mg orally twice weekly. TG02 will be administered on days 1, 4, 8, 11, 15, 18, 22 and 25 of each 28-day cycle (Appendix H). Single agent therapy will continue until disease progression or for up to 12 cycles. Upon completion of 12 cycles without disease progression or unacceptable toxicity, patients may continue on TG02 as determined by the Investigator. The lowest permitted dose will be 100 mg TG02 twice weekly.
Period: Overall Study
Arm/Group | Group A - TG02 + Radiotherapy (RT) Dose 1 100 mg | Group A - TG02 + Radiotherapy (RT) Dose 2 150 mg | Group B - TG02 + Temozolomide (TMZ) Dose 1 100 mg | Group B - TG02 + Temozolomide (TMZ) Dose 2 150 mg | Group C - TG02
Started | 3 | 9 | 3 | 6 | 50
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 9 | 3 | 6 | 50
Not completed — Lack of Efficacy | 2 | 6 | 3 | 4 | 42
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 3
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 3
Not completed — Start of a new anti-cancer treatment | 0 | 0 | 0 | 0 | 1
Not completed — Treatment ongoing | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: In Group A - TG02 + RT - 100 mg, we included patients who received the initial 100 mg TG02 dose. In Group A - TG02 + RT - 150 mg, we included patients who received the initial 150 mg TG02 dose. Similarly, in Group B - TG02 + TMZ -100 mg, we included patients treated at the starting TG02 dose of 100 mg. In Group B - TG02 + TMZ -150 mg, we included patients treated at the starting TG02 dose of 150 mg. In group C we included patients who received the initial TG02 dose of 150 mg.
Groups:
- Group A - TG02 + RT - 100 mg; Group A - TG02 + RT - 150 mg: Newly-diagnosed elderly patients (≥65 years) with IDH1R132H-non mutant and MGMT promoter-unmethylated brain tumors received TG02 orally twice weekly with radiation therapy (RT). TG02 was given on specific days of a 28-day cycle, and RT was administered at 40 Gy over 3 weeks. After combination therapy, patients received maintenance TG02 for up to 12 cycles or until disease progression. The dose of TG02 was escalated from 100 mg to 150 mg based on the occurrence of dose-limiting toxicities (DLTs) in cohorts of patients. If no or only one patient experienced a DLT at 150 mg, it was considered the maximum tolerated dose (MTD). If more than one patient experienced a DLT at either dose, the arm was closed. Patients without DLTs continued at the same dose unless severe side effects required adjustments.
  For the determination of the MTD, patients from Group A - TG02 + Radiotherapy (RT) Dose 1 100 mg and Group A - TG02 + Radiotherapy (RT) Dose 2 150 mg were combined into Group A - TG02 + RT. DLTs of both dose levels were evaluated according to the above and MTD was determined
- Group B - TG02 + TMZ - 100 mg; Group B - TG02 + TMZ - 150 mg: Newly diagnosed elderly patients with IDH1R132H-non-mutant and MGMT promoter-methylated anaplastic astrocytoma or glioblastoma will receive TG02 and temozolomide. TG02 will be administered orally twice weekly in combination with TMZ at a standard 28-day cycle regimen (200 mg/m2) for 5 days. The initial dose of TG02 will be 100 mg, and dose escalation to 150 mg may occur if the dose decision criteria are met.
  For the determination of the MTD, patients from Group B - TG02 + Temozolomide (TMZ) Dose 1 100 mg and Group B - TG02 + Temozolomide (TMZ) Dose 2 150 mg were combined into Group B - TG02 + TMZ. DLTs of both dose levels were evaluated according to the above and MTD was determined
- Group C - TG02: Patients with IDH1R132H-non-mutant anaplastic astrocytoma or glioblastoma at first relapse post TMZ/RT --> TMZ therapy will receive TG02 as a single agent. TG02 will be administered orally twice weekly at an initial dose of 150 mg. Dose adjustments will be made based on tolerability.
  MTD was not an endpoint for this Group
- Total: Total of all reporting groups
Arm/Group | Group A - TG02 + RT - 100 mg | Group A - TG02 + RT - 150 mg | Group B - TG02 + TMZ - 100 mg | Group B - TG02 + TMZ - 150 mg | Group C - TG02 | Total
Number analyzed (Participants) | 3 | 9 | 3 | 6 | 50 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 42 | 42
  >=65 years | 3 | 9 | 3 | 6 | 8 | 29
Age, Continuous [Median (Full Range); unit: years] | 70 [68 to 78] | 73 [70 to 79] | 74 [73 to 77] | 76 [67 to 85] | 57 [19 to 75] | 62.2 [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 5 | 10 | 21
  Male | 2 | 5 | 2 | 1 | 40 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 0 | 0 | 0 | 2 | 2
  Netherlands | 0 | 0 | 0 | 0 | 17 | 17
  France | 2 | 3 | 3 | 4 | 20 | 32
  Switzerland | 1 | 1 | 0 | 0 | 5 | 7
  Germany | 0 | 5 | 0 | 2 | 6 | 13
Karnofsky performance status [Count of Participants; unit: Participants]
  Ambulatory (60) | 0 | 0 | 1 | 0 | 7 | 8
  Cares for one self (70) | 0 | 1 | 2 | 1 | 10 | 14
  Normal activity with effort (80) | 1 | 4 | 0 | 4 | 14 | 23
  Able to carry on normal activities (90) | 2 | 3 | 0 | 1 | 11 | 17
  Normal (100) | 0 | 1 | 0 | 0 | 8 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The primary objective in Groups A and B of the EORTC-1608 study is to establish the Maximum Tolerated Dose (MTD) of TG02 and the recommended phase II dose when combined with either radiotherapy (Group A) or temozolomide (Group B) for glioblastoma treatment. The MTD is the highest dose where no more than one of six patients experiences a Dose Limiting Toxicity (DLT). The study requires a 75% dose intensity for TG02 and the concurrent treatment. The trial uses a two-cohort design to assess TG02 with hypofractionated radiotherapy in patients with an unmethylated MGMT promoter or with temozolomide in those with a methylated promoter. Dose escalation begins at 100 mg TG02 twice weekly. If no DLTs occur in the first three patients, the dose increases to 150 mg. If one patient has a DLT, three more are enrolled at the same dose. If no further DLTs occur, escalation continues. If more than one patient has a DLT, escalation stops, and the previous dose is the MTD.
Time Frame: From the initiation of TG02 treatment until the determination of the Maximum Tolerated Dose (MTD) for each participant, which is expected to occur within the first 28-day cycle for most participants.
Population: Group A - TG02 + radiotherapy (RT) is combining patients from Group A - TG02 + Radiotherapy (RT) Dose 1 who received TG02 at 100 mg and patients from Group A - TG02 + Radiotherapy (RT) Dose 2 who received TG02 at 150 mg.Similarly, Group B - TG02 + TMZ is combining patient from Group B - TG02 + Temozolomide (TMZ) Dose 1 100 mg who received TG02 at 100 mg and patients from Group B - TG02 + Temozolomide (TMZ) Dose 2 who received TG02 at 150 mg.
Measure: Number; unit: mg
Groups:
- Group A - TG02 + Radiotherapy (RT): Newly-diagnosed Elderly patients with Isocitrate dehydrogenase 1 (IDH1) gene non-mutant (IDH1R132H) and MGMT promoter-unmethylated anaplastic astrocytoma or glioblastoma will receive TG02 and radiation therapy. TG02 will be administered orally twice weekly in combination with standard involved-field hypofractionated RT at 39.9 Gy in 15 fractions of 2.66 Gy for 3 weeks. The initial dose of TG02 will be 100 mg, and dose escalation to 150 mg may occur if the dose decision criteria are met.
- Group B - TG02 + Temozolomide (TMZ): Newly diagnosed Elderly patients with IDH1R132H-non-mutant and MGMT promoter-methylated anaplastic astrocytoma or glioblastoma will receive TG02 and temozolomide. TG02 will be administered orally twice weekly in combination with TMZ at a standard 28-day cycle regimen (200 mg/m2) for 5 days. The initial dose of TG02 will be 100 mg, and dose escalation to 150 mg may occur if the dose decision criteria are met.
Arm/Group | Group A - TG02 + Radiotherapy (RT) | Group B - TG02 + Temozolomide (TMZ)
Number analyzed (Participants) | 12 | 9
mg | 150 | 150

2. Primary Outcome: Percentage of Participants Maintaining Progression-free Survival at 6 Months (PFS-6)
Description: The primary endpoint for Group C is Progression-free survival at 6 months (PFS-6), assessed by Response Assessment in Neuro-Oncology (RANO) criteria. Complete Response (CR) is defined as the disappearance of all enhancing measurable and nonmeasurable disease for at least 4 weeks. Partial Response (PR) requires at least a 50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions for at least 4 weeks. Stable Disease (SD) is when the patient does not qualify for CR, PR, or progression, with stable nonenhancing lesions on the same or lower dose of corticosteroids. Progression (PD) is defined as at least a 25% increase in the sum of products of perpendicular diameters of enhancing lesions compared to the smallest measurement at baseline or best response, a significant increase in T2/FLAIR lesion, any new lesion, or clear clinical deterioration not attributable to other causes.
Time Frame: The time frame for assessing PFS spans from the date of consent to either disease progression or death. Data are specifically presented for the 6-month time point.
Population: Analyses are performed in the first 45 patients included in the efficacy population defined as all patients who are eligible and have started their allocated treatment. Due to small sample size, in Group A , we combined patients who received either the initial 100 mg dose or the escalated 150 mg dose and in Group B,we combined patients treated at both the starting dose of 100 mg and the increased dose of 150 mg.In group C we included patients who received the initial dose of 150 mg.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Group C - TG02: Patients with IDH1R132H-non-mutant anaplastic astrocytoma or glioblastoma at first relapse post TMZ/RT --> TMZ therapy will receive TG02 as a single agent. TG02 will be administered orally twice weekly at an initial dose of 150 mg. Dose adjustments will be made based on tolerability.
Arm/Group | Group C - TG02
Number analyzed (Participants) | 45
percentage of participants | 6.7 [2.5 to 14.3]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is a secondary endpoint for Group C. PFS is defined as the number of days from consent to the date of earliest disease progression based on Response Assessment in Neuro Oncology (RANO) criteria (as determined by the Investigator) or to the date of death, if disease progression does not occur. For all groups, the median PFS will be determined. PFS is measured from the start of treatment until the date of disease progression or death, whichever occurs first. Patients without progression or death will be censored at the last date documented to be alive and progression-free.
Time Frame: The time frame for assessing PFS is the duration from the date of consent until disease progression or death. PFS was assessed by its median the point time at which 50% of the patients have experienced death.
Population: Analyses are performed in the efficacy population defined as all patients who are eligible and have started their allocated treatment. In Group A patients received either the initial 100 mg dose or the escalated 150 mg dose and in Group B, patients received the starting dose of 100 mg and the increased dose of 150 mg.In group C we included patients who received the initial dose of 150 mg.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Group A - TG02 + RT - 100 mg: In Group A - TG02 + RT - 100 mg, we included patients who received TG02 at the initial 100 mg dose
- Group A - TG02 + RT - 150 mg: In Group A - TG02 + RT, we included patients who received TG02 at the initial 150 mg dose
- Group B - TG02 + TMZ - 100 mg: In Group B - TG02 + TMZ - 100 mg, we included patients who received TG02 at the initial 100 mg dose
- Group B - TG02 + TMZ - 150 mg: In Group B - TG02 + TMZ - 150 mg, we included patients who TG02 received at the initial 100 mg dose
- Group C - TG02: In Group C - TG02 , we included patients who received TG02 at the initial 150 mg dose
Arm/Group | Group A - TG02 + RT - 100 mg | Group A - TG02 + RT - 150 mg | Group B - TG02 + TMZ - 100 mg | Group B - TG02 + TMZ - 150 mg | Group C - TG02
Number analyzed (Participants) | 3 | 9 | 3 | 6 | 46
Months | 2.4 [1.8 to 2.4] | 4.4 [1.4 to 6.7] | 4.9 [2.6 to 4.9] | 7.1 [4.6 to 7.1] | 1.87 [1.64 to 1.94]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is a secondary endpoint for Group C. OS is defined as the number of days from consent to the date of death due to any cause. If a patient has not died, the data was censored at the last date documented to be alive. For all groups, the median OS was determined. The median OS was extracted from the Kaplan-Meier OS curve,
Time Frame: The time frame for assessing OS is from consent to the date until death or the end of the study, whichever comes first. OS was assessed by its median the point time at which 50% of the patients have experienced death.
Population: The intent-to-treat (ITT) population was used which is defined as all enrolled patients who will be analyzed in the arm they were allocated by randomization. In Group A patients received either the initial 100 mg dose or the escalated 150 mg dose and in Group B, patients received the starting dose of 100 mg and the increased dose of 150 mg.In group C we included patients who received the initial dose of 150 mg.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Group A - TG02 + RT - 150 mg: In Group A - TG02 + RT - 150 mg, we included patients who received TG02 at the initial 150 mg dose
- Group B - TG02 + TMZ - 150 mg: In Group B - TG02 + TMZ - 150 mg, we included patients who received TG02 at the initial 150 mg dose
Arm/Group | Group A - TG02 + RT - 100 mg | Group A - TG02 + RT - 150 mg | Group B - TG02 + TMZ - 100 mg | Group B - TG02 + TMZ - 150 mg | Group C - TG02
Number analyzed (Participants) | 3 | 9 | 3 | 6 | 50
Months | 9.3 [1.8 to 9.3] | 6.7 [4.4 to 6.7] | 14.6 [6.3 to 14.6] | 11.3 [5.6 to 11.3] | 7.00 [4.90 to 8.84]

5. Secondary Outcome: Objective Response
Description: Objective Response (OR) is a secondary endpoint for Group C. For patients with measurable disease after debulking or non-surgical patients with measurable disease after surgery for recurrence, the best overall response distribution (BOR), objective response rate (PR+CR), complete response rate, and duration of response (DOR) was assessed. The objective response rate is the proportion of patients who achieve a partial response (PR) or complete response (CR), while the complete response rate is the proportion of patients who achieve a CR. The duration of response (DOR) is the time from the first documented response (PR or CR) to the date of disease progression or death, whichever occurs first.
Time Frame: Time frame for assessing response is from the initiation of treatment with TG02 until disease progression or death. It was not assessed at specific time point but throughout the study. The OR rate is determined based on the best response observed.
Population: Analysis population is the intent-to-treat (ITT) population defined as all enrolled patients who will be analyzed in the arm they were allocated by randomization. In Group A patients received either the initial 100 mg dose or the escalated 150 mg dose and in Group B, patients received the starting dose of 100 mg and the increased dose of 150 mg.In group C we included patients who received the initial dose of 150 mg.
Measure: Number; unit: Number of participants
Arm/Group | Group A - TG02 + RT - 100 mg | Group A - TG02 + RT - 150 mg | Group B - TG02 + TMZ - 100 mg | Group B - TG02 + TMZ - 150 mg | Group C - TG02
Number analyzed (Participants) | 3 | 9 | 3 | 6 | 50
Number of participants | 0 | 0 | 0 | 3 | 1

6. Secondary Outcome: Neurological Progression-free Survival
Description: Neurological progression-free survival (NPFS) is a secondary endpoint for Group C. NPFS is defined based on the Neurologic Assessment in Neuro-Oncology (NANO) criteria. NPFS is measured from the date of enrollment in the trial until the date of first neurological progression or death, whichever occurs first. If a patient does not experience neurological progression or death, the data will be censored at the last date of post-baseline neurological assessment. The median NPFS will be determined.
Time Frame: The time frame for assessing NPFS spans from the date of consent to either disease progression or death.NPFS was assessed by its median the point time at which 50% of the patients have experienced death.
Population: Analyses are performed in the efficacy population defined as all patients who are eligible and have started their allocated treatment (at least one study drug dose). In Group A patients received either the initial 100 mg dose or the escalated 150 mg dose and in Group B, patients received the starting dose of 100 mg and the increased dose of 150 mg.In group C we included patients who received the initial dose of 150 mg.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Group B - TG02 + TMZ - 150 mg: In Group B - TG02 + RT - 150 mg, we included patients who received TG02 at the initial 150 mg dose
Arm/Group | Group A - TG02 + RT - 100 mg | Group A - TG02 + RT - 150 mg | Group B - TG02 + TMZ - 100 mg | Group B - TG02 + TMZ - 150 mg | Group C - TG02
Number analyzed (Participants) | 3 | 9 | 3 | 6 | 46
Months | 8.4 [1.8 to 8.4] | 6.5 [1.6 to 8.1] | 14.6 [2.60 to 14.6] | 11.3 [4.6 to 11.3] | 2.27 [1.87 to 4.73]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and All-Cause Mortality evaluated from TG02 treatment start to 30 days post-final dose or until chronic/stable. SAEs/serious suspected adverse reactions reported within 30 days followed until resolved/chronic/stable. All-Cause Mortality assessed until study end or loss to follow-up. Adverse Events (AEs) and All-Cause Mortality were evaluated up to 25 months from start of enrolment.
Description: Both serious adverse events (SAEs) and non-serious AEs were collected. We reported SAEs and all AEs. Non serious AEs are accounted for in the all AEs report. All AEs report is included in the Other (Not Including Serious) section. All-cause mortality was assessed all registered patients. SAEs and all AEs were assessed in the registered patients who have started their allocated treatments.
Arm/Group | Group A - TG02 + RT - 100 mg | Group A - TG02 + RT - 150 mg | Group B - TG02 + TMZ - 100 mg | Group B - TG02 + TMZ - 150 mg | Group C - TG02
All-Cause Mortality (participants affected / at risk) | 3/3 | 7/9 | 3/3 | 3/6 | 42/50
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/9 | 0/3 | 3/6 | 13/50
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 3/3 | 6/6 | 46/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - TG02 + RT - 100 mg (N=3) | Group A - TG02 + RT - 150 mg (N=9) | Group B - TG02 + TMZ - 100 mg (N=3) | Group B - TG02 + TMZ - 150 mg (N=6) | Group C - TG02 (N=50)
Colonic Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Clinical Status Worsening (General disorders) | 0 | 0 | 0 | 0 | 1
Other AE (General disorders) | 0 | 1 | 0 | 0 | 0
Worsening Of General Condition (General disorders) | 0 | 1 | 0 | 0 | 0
Worsening Of General Condition Due To Clinical Progression (General disorders) | 0 | 0 | 0 | 0 | 1
Dystelectasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Inhalation Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Brain Edema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Convulsive Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Edema Cerebral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neurological Worsening (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Other AE* (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Right Capsulolenticular Intraparenchymal Hematomas And Oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 2 | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Worsening Of Hemiparesis Left (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Skin Rash Toxidermia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Pulmonary Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - TG02 + RT - 100 mg (N=3) | Group A - TG02 + RT - 150 mg (N=9) | Group B - TG02 + TMZ - 100 mg (N=3) | Group B - TG02 + TMZ - 150 mg (N=6) | Group C - TG02 (N=50)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 1 | 0 | 0 | 1 | 0
Hemianopsie Left (Eye disorders) | 0 | 1 | 0 | 0 | 0
Periorbital Edema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Colonic Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 13
Diarrhea (Gastrointestinal disorders) | 1 | 5 | 2 | 5 | 20
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Fecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gallstone Without Cholecystitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 1 | 4 | 19
Pain Hypochondrial Left (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0 | 4 | 9
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 3
Balance Disorder (General disorders) | 0 | 0 | 0 | 1 | 0
Clinical Status Worsening (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 4 | 3 | 3 | 20
Fever (General disorders) | 0 | 2 | 0 | 2 | 2
Flu Like Symptoms (General disorders) | 0 | 0 | 0 | 0 | 1
Gait Disturbance (General disorders) | 0 | 1 | 0 | 1 | 1
Ideomotor Deceleration (General disorders) | 0 | 0 | 0 | 0 | 1
Loss Of Appetite (General disorders) | 0 | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Other AE (General disorders) | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pain In Both Feet (General disorders) | 1 | 0 | 0 | 0 | 0
Pain Shoulder (General disorders) | 0 | 0 | 0 | 0 | 1
Reduced General Condition (General disorders) | 0 | 1 | 0 | 0 | 0
Transient Hemiparesis Left Side (General disorders) | 0 | 1 | 0 | 0 | 0
Worsening Of General Condition (General disorders) | 0 | 1 | 0 | 1 | 0
Worsening Of General Condition Due To Clinical Progr (General disorders) | 0 | 0 | 0 | 0 | 1
Allergic Reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Bronchial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Covid-19 Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dystelectasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes Simplex Reactivation (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Inhalation Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 3 | 7
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 1 | 2
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Cardiac Troponin T Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Cd4 Lymphocytes Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Cpk Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased Lymphocyte Count (Investigations) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Investigations) | 0 | 0 | 0 | 1 | 0
Hyponatremia (Investigations) | 0 | 1 | 0 | 0 | 0
Increased Alt (Investigations) | 0 | 0 | 0 | 0 | 1
Increased Crp (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 2 | 1 | 4 | 12
Neutropenia (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 3 | 6
Platelet Count Decreased (Investigations) | 0 | 0 | 1 | 2 | 3
Weight Gain (Investigations) | 0 | 0 | 0 | 0 | 1
Weight Loss (Investigations) | 0 | 1 | 0 | 0 | 2
White Blood Cell Decreased (Investigations) | 0 | 1 | 0 | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoproteinemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Thigh Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neoplasm Benign, Malignant And Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Aphasia (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Brain Edema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral Edema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cognitive Disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Convulsive Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Edema Cerebral (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Frontal Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 15
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hemiparesis Left (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischemia Cerebrovascular (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Left Hemiparisis 3/5 (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Left Lower Limb Deficit (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Motor Degradation In The Left Hand (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Muscle Weakness Left Sided (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Muscle Weakness Left-Sided (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Muscle Weakness Right-Sided (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Neurological Worsening (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Other Nervous System Disorders- Hemiparesis Right (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Right Capsulolenticular Intraparenchymal Hematomas A (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 3 | 2 | 1 | 8
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Worsening Of Hemiparesis Left (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Worsening Of Neurocognitive Deficits (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary Frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Common Cold (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Bedsore (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin And Subcutaneous Tissue Disorders, Other: Wound (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin Rash Toxidermia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Hematoma (Vascular disorders) | 1 | 0 | 1 | 1 | 1
Hot Flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 0 | 0 | 1 | 3
Vascular Access Compilation (Vascular disorders) | 0 | 0 | 0 | 1 | 0 — Vascular Access Compilation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03224104/Prot_SAP_000.pdf